CLINICAL TRIAL: NCT03419793
Title: Effect of Segmental Muscle Vibration on Upper Extremity Functional Ability Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Annino, Principal Investigator, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 212/17
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy intervention and segmental muscle vibration (Experimental): physiotherapy intervention and segmental muscle vibration device
  Interventions: Device: segmental vibration device; Other: physical therapy exercises
- physical therapy intervention (Sham Comparator): physical therapy intervention alone
  Interventions: Other: physical therapy exercises

INTERVENTIONS:
Device: segmental vibration device — segmental vibration device
  Other Names: physical therapy intervention
  Arms: physical therapy intervention and segmental muscle vibration
Other: physical therapy exercises
  Other Names: manual resistance exercise

SUMMARY:
Background and objective: Upper extremity functional impairments are common consequences post stroke. The aim of this study was to investigate the influence of Segmental muscle vibration (SMV) application along with supervised physical therapy (SPT) on improving activities of daily living (ADL) and motor recovery on the hemiparetic upper extremity in patients with stroke.

Methods: A sample of 37 patients post stroke (29 males) was randomly assigned to either supervised physical therapy (SPT) control group (n=18) or supervised physical therapy and segmental muscle vibration (SPT-SMV) experimental group (n=19). All patients received 3 sessions per week of SPT for 8 weeks. The SPT-SMV experimental group received SMV at the end of each SPT session. Outcome measures used were Barthel Index (BI), Modified Ashworth Scale (MAS), Manual Muscle Testing (MMT), and goniometry for Range of Motion (ROM) assessment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stroke

Exclusion Criteria:

* if they had any serious orthopedic injury/disease, cardiopulmonary problems or suffered from a neurological disease (other than stroke).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
goniometry | Change from Baseline Range of Motion at 8 weeks
  Range of motion assessed by goniometry; is the measurement of angles, particularly those formed by joints. These angles may be measured in a standing position or in flexion or extension.

SECONDARY OUTCOMES:
Barthel Index (BI) | Change from Baseline Functional level at 8 weeks
  The Barthel Index of Activities of Daily Living (BI). Measure of functional disability. The BI consisting of 10 common activities of daily living (ADL) activities, administered through direct observation. These are assessed for independence/ dependence and scored via an arbitrary weighting system (originally applied to reflect nursing care and social acceptability). Eight of the ten items represent activities related to personal care; the remaining 2 are related to mobility. The index yields a total score out of 100 - the higher the score, the greater the degree of functional independence
Manual Muscle Testing (MMT) | Change from Baseline Muscle power at 8 weeks
  Muscle strength assessed by using manual muscle testing (MMT) . The six- point Medical Research Council (MRC) Scale is the most often used system, with the procedures detecting the magnitude of strength by grading muscle strength from 0 to 5. In which a score of 0 was no contraction, 1 was a flicker of contraction, 2 was active movement with gravity eliminated, 3 was active movement against gravity, 4 was active movement against gravity and resistance and 5 was normal power
Modified Ashworth Scale (MAS) | Change from Baseline muscle tone at 8 weeks
  The scale is used to assign a subjective rating of the amount of resistance or tone perceived by the examiner as a limb is moved through its full range of motion. The original Ashworth scale consisted of 5 grades from 0 - 4. in which score of 0 was no increase in muscle tone, 1 was Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension, 1+ was slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM, 2 was more marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3 was considerable increase in muscle tone, passive movement difficult and 4 was affected part(s) rigid in flexion or extension

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Annino, PhD, Study Director — department of medicine systems